CLINICAL TRIAL: NCT05742932
Title: Prospective Study to Evaluate the Performance and the Safety of Global D's Implants of Craniomaxillofacial Surgery (CMF) Ranges Indicated for Trauma Surgery (CMF-TRAUMA)
Status: Active, not recruiting | Type: Observational
Sponsor: Global D (Industry)
Responsible Party: Sponsor
Other Study IDs: 2102-G-CMF-TRAUMA-R
Record Dates: First submitted 2023-02-15; First posted 2023-02-24 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Trauma Injury; Maxilla Fracture; Maxillofacial Trauma
Keywords: Performance; Safety; Screw; Plate; Medical device; Trauma surgery; Cranio-maxillofacial; Global D
MeSH Terms: conditions — Accidental Injuries; Maxillary Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Male and female, major or minor patients. The patients have maxillary, mandibular, maxillomandibular fracture with/without annex face or skull fracture, and will be treated by trauma surgery.
  Interventions: Device: Trauma surgery using Global D's implants.

INTERVENTIONS:
Device: Trauma surgery using Global D's implants. — Major or minor participants who will be treated by an trauma surgery with ORTRAUTEK® or MINITEK/MICROTEK® implant(s).

SUMMARY:
This study is set up within the framework of the European Union regulation 2017/745 on medical devices. Its objective is to confirm the performance and safety of the Global D implants (ORTRAUTEK® and MINITEK/MICROTEK®) used for trauma surgery.

DETAILED DESCRIPTION:
Study design : Non-interventional, prospective, multicentric, national, open-label, non-comparative study.

Investigators : 5 sites in France.

A statistical evaluation will be performed on those data in order to determine the performance and the security of those devices.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient, major or minor (11 years old minimum)
* Patient undergoing surgery on the mandible and/or maxilla (mandatory), with or without associated facial fractures (orbit, upper two-thirds of the face, skull)
* Patient with abilities to read, understand and answer to the study questionnaires.
* Patient (and his legal representative if minor) who signed the study consent form.
* Patient affiliated to a social security system.

Exclusion Criteria:

* Patient allergic to one of the components of the implants
* Patient with physical or mental inabilities that will compromise the follow-up during the study
* Patient with acute or chronic infection (local or systemic)
* Patients with bone's tumors in the anchorage area of the implant
* Person on legal protection
* Pregnant or breastfeeding women

Min Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population is composed of male and female, major or minor, who will be treated by trauma surgery. The patients will have maxillary, mandibular or maxillomandibular fractures with/without annex skull's or face's fractures.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Performance of the Global D's implants used for trauma surgery assessed by the evaluation of the functional jaw activity 6 months after the surgery | 6 months
  The functional jaw activity will be evaluated with the Mandibular Function Impairment Questionnaire (MFIQ) 6 months after the surgery. This questionnaire have 17 items, that have to be answered with a Likert scale from 1 (No problem) to 5 (very hard or impossible).

SECONDARY OUTCOMES:
Performance of the Global D implants used for trauma surgery - Outcome Measure 1 | 6 months
  Evolution of functional jaw activity, assessed by the evolution of MFIQ questionnaire's answers at 3 timepoints (pre-operative, 4-6 weeks after the surgery and 6 months after the surgery). The post-operatives answers will be compared to the pre-operative answers.
Security of the Global D implants used for trauma surgery - Outcome Measure 2 | 1 year
  Adverse events identification, assessment and follow-up.
Security of the Global D implants used for trauma surgery - Outcome Measure 3 | 6 months
  Bone consolidation after the surgery, 4-6 weeks after the surgery and 6 months after the surgery.
Performance of the Global D implants used for trauma surgery - Outcome Measure 4 | 6 months
  Evolution of the patient's buccal quality of life in preoperative, 4-6 weeks after the surgery and 6 months after the surgery. To assessed this buccal quality of life, the patient will answered to Oral Health Impact Profile (OHIP-14) questionnaire. This questionnaire is composed of 14 questions, the patient can answer from 0 (Never) to 4 (Very Often).
Surgeon satisfaction on the implant's utilisation - Outcome Measure 5 | Immediately following surgery
  Assessment by a satisfaction questionnaire, specially developed for the study, completed by the surgeon after the surgery. The surgeon evaluates each item using a likert scale (Highly Satisfied/ Satisfied/ Unsatisfied/Very Unsatisfied)
Localisation and annex fractures data collection | 12 months
  If applicable, localisation and annex fractures data collection, and the medical device's references used to treat thoses fractures.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Chauvel-Picard, MD, Principal Investigator — Cranio-maxillofacial surgeon
Locations (2):
- France (2):
  - Hopital de la Croix Rousse - Hospices Civils de Lyon (FRANCE), Lyon
  - Hopital Femme Mère Enfant - Hospices Civils de Lyon (FRANCE), Lyon